CLINICAL TRIAL: NCT05320939
Title: Immunological Basis for Mepolizumab Activity in COPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Temple University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISS Proposal # 12342
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: A pilot open-label single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mepolizumab 100mg (Experimental): The Investigators will recruit a total of 30 subjects for this study (all subjects for the mepolizumab treatment).
  Interventions: Drug: Mepolizumab 100 MG

INTERVENTIONS:
Drug: Mepolizumab 100 MG — 30 subjects (≥ 300 eosinophils/ul) will receive mepolizumab 100 mg subcutaneously every 4 weeks for 5 complete doses.

SUMMARY:
The current literature suggests that the mode of action of mepolizumab is to bind with Interleukin (IL)-5 and block the interaction of IL-5 with the IL-5Ra receptor on eosinophils. This removal of IL-5 may not explain all of the effects of mepolizumab. The investigators propose a set of studies to systematically examine the spectrum of effects of this drug on the immune system.

DETAILED DESCRIPTION:
The investigators will recruit a total of 30 Chronic Obstructive Pulmonary Disease (COPD) participants from the Temple University Hospital Lung Center Clinic. All participants will have moderate to severe COPD and have a history of 2 or more acute exacerbations in the past year, and eosinophil counts of greater than 300 cells/ul. The investigators studies will include an analysis of the status of the systemic and lung inflammatory phenotype of the major leukocyte populations, using multiparameter flow cytometry. The investigators will couple these studies with an analysis of a panel of inflammatory and anti-inflammatory biomarkers in both the blood and bronchoalveolar lavage fluid. Very importantly, the investigators will characterize the functional capacity of T cells, B cells, monocytes, and granulocytes during drug therapy. By using this approach, the investigators believe a more complete understanding of the scope of activity of mepolizumab at the level of immune competence will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral blood eosinophil count of ≥300 cells/μL from the hematology sample collected and a documented historical blood eosinophil count of ≥300/μL in the 12 months prior.
* Clinically documented history of Chronic Obstructive Pulmonary Disease (COPD) for at least 1 year in accordance with the definition by the American Thoracic Society/European Respiratory Society. A measured pre-and post-salbutamol FEV1/FVC ratio of <0.70.
* Well-documented history (e.g., medical record verification) in the 12 months prior which includes 2 or more moderate COPD exacerbations that were treated with systemic corticosteroids (intramuscular (IM), intravenous, or oral) with or without antibiotics OR at least one severe COPD exacerbation requiring hospitalization.
* Current or former cigarette smokers with a history of cigarette smoking of ≥10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior.
* A female is eligible if the participant is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP) or 2) Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1% during the intervention period and for at least 16 weeks after the last dose of study intervention.
* A WOCBP must have a negative highly sensitive pregnancy urine test within 24 hours before the first dose of study intervention.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Past history or concurrent diagnosis of asthma.
* An α1-antitrypsin deficiency as the underlying cause of COPD are excluded.
* Active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Pneumonia, COPD exacerbation, or lower respiratory tract infection within prior 4 weeks.
* Lung volume reduction surgery within the last 12 months.
* Participating in acute phase of a pulmonary rehabilitation program within last 4 weeks.
* Receiving treatment with oxygen more than 2 Liters(L)/minute at rest over 24 hours. If receiving oxygen treatment, an oxyhemoglobin saturation (as measured by PulseOx) greater than or equal to 89% while breathing supplemental oxygen.
* Myocardial infarction or unstable angina in the prior 6 months.
* Unstable or life threatening cardiac arrhythmia requiring intervention in the prior 3 months.
* New York Heart Association (NYHA) Class IV Heart failure.
* Historical or current evidence of clinically significant, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled.
* Other conditions that could lead to elevated eosinophils such as Hypereosinophilic syndromes including Eosinophilic Granulomatosis with Polyangiitis, or Eosinophilic Esophagitis.
* A known pre-existing parasitic infestation within prior 6 months.
* A current malignancy or previous history of cancer in remission for less than 12 months.
* A known immunodeficiency (e.g. human immunodeficiency virus - HIV), other than that explained by the use of corticosteroids taken for COPD.
* Cirrhosis or current unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice. Stable noncirrhotic chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C -e.g., presence of hepatitis B surface antigen [HbsAg] or positive hepatitis C antibody test result) is acceptable if the participant otherwise meets entry criteria.
* Received interventional product in previous mepolizumab studies.
* Received any monoclonal antibody within 5 half-lives.
* Received an investigational drug within prior 30 days or within 5 drug half-lives of the investigational drug, whichever is longer.
* Received short term use of oral corticosteroids within prior 30 days.
* A known allergy or sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator contraindicates participation in the study or intolerance to another monoclonal antibody or biologic including history of anaphylaxis to another biologic.
* Participants with, conditions that will limit the validity of informed consent to participate in the study, e.g uncontrolled psychiatric disease or intellectual deficiency.
* A known or suspected history of alcohol or drug abuse within prior 2 years.
* Is an Investigator, sub-Investigator, study coordinator, employee of a participating Investigator or study site, or immediate family member of the aforementioned that is involved in this study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of peripheral blood eosinophil and B cell levels | 6 months
  Peripheral blood eosinophil and B cell number counts

SECONDARY OUTCOMES:
Change from baseline of peripheral blood T cells | 6 months
  Peripheral blood T cell number counts
Change from baseline of peripheral blood monocytes | 6 months
  Peripheral blood monocyte number counts
Change from baseline of peripheral blood neutrophils | 6 months
  Peripheral blood neutrophil cell number counts
Change from baseline of peripheral blood NK cells | 6 months
  Peripheral blood NK cell number counts
Change from baseline of peripheral blood dendritic cells | 6 months
  Peripheral blood dendritic cell number counts
Change from baseline of peripheral blood CCL11 levels | 6 months
  Blood CCL11 pg/ml
Change from baseline of peripheral blood CCL24 levels | 6 months
  Blood CCL24 pg/ml
Change from baseline of peripheral blood CCL26 levels | 6 months
  Blood CCL26 pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rogers, PhD, Principal Investigator — Temple University